CLINICAL TRIAL: NCT03837639
Title: Effects of Arm-crank Exercise Training on Cardiovascular Function of Patients With Peripheral Artery Disease: a Randomized Controlled Trial
Brief Title: Arm-crank Exercise Training on Cardiovascular Function of Patients With Peripheral Artery Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: University of Nove de Julho (Other); Northumbria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PAD01
Record Dates: First submitted 2019-02-07; First posted 2019-02-12 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Peripheral Arterial Disease; Intermittent Claudication; Hypertension
Keywords: arm-crank; exercise training; cardiovascular function
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Hypertension | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm crank ergometer (Experimental): Arm-crank exercise group will be performed twice a week for 12 weeks. In the first weeks of training, each session will consist of 15 bouts, two active minutes and two minutes of passive interval, consisting of 60 minutes of session (30 minutes of active exercise). After the first three weeks of training, the exercise time will progressively increase by one minute every 3 weeks and the recovery period will be decreased, completing, at the end, a maximum volume of 10 bouts of five minutes of exercise and one minute of passive interval. The intensity of the exercise will be determined by the load equivalent to the range of 13 - 15 of The Borg Rating of Perceived Exertion, considered as somewhat hard to hard.
  Interventions: Other: Arm ergometer
- Treadmill ergometer (Experimental): Walking exercise group will be performed twice a week for 12 weeks. In the first weeks of training, each session will consist of 15 bouts, two active minutes and two minutes of passive interval, consisting of 60 minutes of session (30 minutes of active exercise). After the first three weeks of training, the exercise time will progressively increase by one minute every 3 weeks and the recovery period will be decreased, completing, at the end, a maximum volume of 10 bouts of five minutes of exercise and one minute of passive interval. The intensity of the exercise will be determined by the load equivalent to the range of 13 - 15 of The Borg Rating of Perceived Exertion, considered as somewhat hard to hard.
  Interventions: Other: Treadmill ergometer
- Control group (Other): Patients randomized to control group will attend to meetings with the researcher team twice a week during the 12 weeks. At these meetings, patients will perform manual tasks, with or without the use of artistic materials, cultural programs, cooking classes and home care, without any exercise component. This CG practice will be performed in order to minimize the effects of the patient's bi- weekly commitment and displacement to the training site, to minimize the influence of the patient- researcher contact and also minimize the convivial effect among the patients themselves, which will occur in the other two groups.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Arm ergometer — Arm-crank exercise group will be performed twice a week for 12 weeks. In the first weeks of training, each session will consist of 15 bouts, two active minutes and two minutes of passive interval, consisting of 60 minutes of session (30 minutes of active exercise). After the first three weeks of training, the exercise time will progressively increase by one minute every 3 weeks and the recovery period will be decreased, completing, at the end, a maximum volume of 10 bouts of five minutes of exercise and one minute of passive interval. The intensity of the exercise will be determined by the load equivalent to the range of 13 - 15 of The Borg Rating of Perceived Exertion, considered as somewhat hard to hard
  Arms: Arm crank ergometer
Other: Treadmill ergometer — Walking exercise group will be performed twice a week for 12 weeks. In the first weeks of training, each session will consist of 15 bouts, two active minutes and two minutes of passive interval, consisting of 60 minutes of session (30 minutes of active exercise). After the first three weeks of training, the exercise time will progressively increase by one minute every 3 weeks and the recovery period will be decreased, completing, at the end, a maximum volume of 10 bouts of five minutes of exercise and one minute of passive interval. The intensity of the exercise will be determined by the load equivalent to the range of 13 - 15 of The Borg Rating of Perceived Exertion, considered as somewhat hard to hard.
  Arms: Treadmill ergometer
Other: Control group — Patients randomized to control group will attend to meetings with the researcher team twice a week during the 12 weeks. At these meetings, patients will perform manual tasks, with or without the use of artistic materials, cultural programs, cooking classes and home care, without any exercise component. This CG practice will be performed in order to minimize the effects of the patient's bi- weekly commitment and displacement to the training site, to minimize the influence of the patient- researcher contact and also minimize the convivial effect among the patients themselves, which will occur in the other two groups.
  Arms: Control group

SUMMARY:
The aim of the study is to analyze the effect of 12 weeks of arm crank exercise (ACE) training on cardiovascular function in PAD patients, and compare it with treadmill exercise (TE), the actual recommendation for this patients. In this clinical trial, 45 patients will be allocated randomly in three experimental groups: ACE training, TE and control group. ACE and TE groups will perform exercises twice a week with the intensity equivalent to 13- 15 on Borg's Subjective Perception Exertion Scale. Patients in control group will meet twice a week, however only to perform diverse activities and group living, without any type of exercise involved. All groups will be encouraged to increase their levels of activity, as they are usually guided in medical consultations. Before and after 12 weeks of intervention, cardiovascular function, functional capacity, cognition, and quality of life will be assessed.

DETAILED DESCRIPTION:
Arm-crank exercise (ACT) is an alternative exercise strategy for patients with symptomatic peripheral artery disease (PAD) due the benefits on functional capacity and quality of life, besides provoking less or no pain symptoms during the execution. This study sought to describe the protocol of a study that will analyse the effect of ACT exercise on walking capacity, cardiovascular function, cognition and quality of life in patients with symptomatic PAD.

This is a three-armed randomized, prospective, single-blind data collection, single-center, controlled study enrolling 45 patients with symptomatic PAD which will be randomized into 3 intervention groups: walking training (WT), ACT (WT and AC: 15 to 10 sets of 2 to 5 minutes, Borg 13 to 15) and control group (CG). Before and after 12 weeks of intervention, cardiovascular function (ambulatory blood pressure , clinic blood pressure, central blood pressure, heart rate variability, arterial stiffness, vascular function), functional capacity (six-minute walking test, 2 minute step test [2 MST], Walking impairment questionnaire [WIQ], Walking estimated limitation calculated by history [WELCH], Baltimore activity scale for intermittent claudication, handgrip test and short physical performance battery [SPPB]), cognition (executive function and memory) and quality of life (short version of world health organization quality of life and vascular quality of life questionnaire [VASCUQOL-6]) will be assessed.

This is the first trial to evaluate the effects of ACT on regulatory mechanisms of cardiovascular system in PAD patients. If the results are as expected, they will provide evidence of ACT in promoting cardiovascular benefits in symptomatic PAD population.

ELIGIBILITY:
Inclusion Criteria:

* PAD stage II
* Ankle brachial index <0.90 in one or both lower limbs;
* Women in post-menopause phase without hormone replacement therapy
* Not an active smoker;
* Able to perform exercise training;

Patients selected to participate in the study will be only excluded if:

* Change their medication;
* Present any health impairment that contraindicates the practice of physical exercise during the study;

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-06-10 (Actual); Primary Completion 2022-12-10 (Estimated); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
ambulatory blood pressure | Change from baseline in ambulatory blood pressure at 12 weeks
  Systolic, diastolic and mean blood pressure will be measured before and after 12 weeks of intervention period on intervention and control group by an automatic ambulatory blood pressure monitor (Cardios, São Paulo, Brazil).

SECONDARY OUTCOMES:
Clinic blood pressure | Change from baseline in ambulatory blood pressure at 12 weeks
  Systolic and diastolic brachial blood pressure will be measured before and after 12 weeks of intervention period on intervention and control group by an automatic blood pressure monitor (HEM-742, Omron Healthcare, Japan).
Central blood pressure | Change from baseline in ambulatory blood pressure at 12 weeks
  Systolic and diastolic central blood pressure will be measured before and after 12 weeks of intervention period on intervention and control group by an automatic blood pressure monitor (HEM-742, Omron Healthcare, Japan).
Heart rate variability | Change from baseline in ambulatory blood pressure at 12 weeks
  Heart rate variability will be measured before and after 12 weeks of intervention period on intervention and control group by heart rate monitor (Polar, RS 800, USA).
Arterial stiffness | Change from baseline in arterial stiffness at 12 weeks
  Carotid femoral pulse wave velocity will be measured before and after 12 weeks of intervention period on intervention and control group by pulse wave velocity measurement with applanation tonometry (SphygmoCor, AtCor Medical, Australia).
Vascular function | Change from baseline in flow-mediated vasodilation at 12 weeks
  Flow-meadiated dilation will be measured before and after 12 weeks of intervention period on intervention and control group by a flow mediated dilation measurement with an ultrasound image (HDI 5000 Sono CT, Philips, The Netherlands).
Walking capacity | Change from baseline in walking distance at 12 weeks
  Six-minute walking test will be measured before and after 12 weeks of intervention
March in place | Change from baseline in the number of the steps at 12 weeks
  Two-minute step test will be measured before and after 12 weeks of intervention
Subjective measurement of walking capacity | Change from baseline in the walking impairment questionnaire score after 12 weeks
  Walking impairment questionnaire will be measured before and after 12 weeks of intervention
Subjective measurement of walking capacity compared to healthy subjects | Change from baseline in the Walking estimated limitation calculated by history questionnaire score after 12 weeks
  Walking estimated limitation calculated by history questionnaire will be measured before and after 12 weeks of intervention
Overall strength test | Change from baseline in kgf of the handgrip test after 12 weeks
  Handgrip strength test will be measured before and after 12 weeks of intervention
Symptoms of intermittent claudication | Change from baseline in the Baltimore Activity Scale for Intermittent Claudication score after 12 weeks
  The Baltimore Activity Scale for Intermittent Claudication is a questionnaire that will be measured before and after 12 weeks of intervention.
General functional capacity | Change from baseline in the Short Physical Performance Battery score after 12 weeks
  The Short Physical Performance Battery will be measured before and after 12 weeks of intervention.
Specific quality of life of vascular patients | Change from baseline in the Vascular quality of life questionnaire score after 12 weeks
  The Vascular quality of life questionnaire will be measured before and after 12 weeks of intervention.
General quality of life | Change from baseline in the World Health Organization Quality of Life score after 12 weeks
  The World Health Organization Quality of Life questionnaire will be measured before and after 12 weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Hélcio Kanegusuku, PhD, Study Chair — Israelite Institute for Education and Research
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
We are planing to share our data in the future.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication of the main paper.
Access Criteria: Ask to authors permision.

REFERENCES:
- [Background] Cavalcante BR, Ritti-Dias RM, Soares AH, Lima AH, Correia MA, De Matos LD, Gobbi F, Leicht AS, Wolosker N, Cucato GG. A Single Bout of Arm-crank Exercise Promotes Positive Emotions and Post-Exercise Hypotension in Patients with Symptomatic Peripheral Artery Disease. Eur J Vasc Endovasc Surg. 2017 Feb;53(2):223-228. doi: 10.1016/j.ejvs.2016.11.021. Epub 2016 Dec 21. PMID 28012910
- [Derived] Costa RM, Kanegusuku H, Cucato GG, Wolosker N, Ritti-Dias RM, Correia MA. Arm Crank Exercise Training Improves Ambulatory Blood Pressure in Patients With Symptomatic Peripheral Artery Disease: Randomized Controlled Trial. J Cardiopulm Rehabil Prev. 2024 Mar 1;44(2):145-147. doi: 10.1097/HCR.0000000000000829. Epub 2023 Nov 30. No abstract available. PMID 38032247
- [Derived] Jansen SC, Abaraogu UO, Lauret GJ, Fakhry F, Fokkenrood HJ, Teijink JA. Modes of exercise training for intermittent claudication. Cochrane Database Syst Rev. 2020 Aug 20;8(8):CD009638. doi: 10.1002/14651858.CD009638.pub3. PMID 32829481